CLINICAL TRIAL: NCT03264157
Title: A Prospective, Randomized, Double-Blind Parallel-group, Non-inferiority Phase II/III Study of the Safety and Effectiveness of BPL HRIG With Co Administration of Active Rabies Vaccine in Healthy Subjects
Brief Title: Safety and Effectiveness of BPL HRIG With Active Rabies Vaccine in Healthy Subjects
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Bio Products Laboratory (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RIG01
Record Dates: First submitted 2017-08-22; First posted 2017-08-29 (Actual); Results first posted 2020-02-11 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-01

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Treatment A: BPL HRIG + active rabies vaccine Treatment B: Comparator HRIG + active rabies vaccine
Who Masked: Participant, Investigator
Masking Description: Double-blind study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BPL HRIG + RabAvert (Experimental): 20 IU/kg dose HRIG + active rabies vaccine
  Interventions: Drug: HRIG; Biological: RabAvert
- Comparator HyperRab + RabAvert (Active Comparator): 20 IU/kg dose HRIG + active rabies vaccine
  Interventions: Drug: HyperRAB; Biological: RabAvert

INTERVENTIONS:
Drug: HRIG — A 20 IU/kg dose of BPL HRIG will be given on Day 0 via IM injection.
  Arms: BPL HRIG + RabAvert
Drug: HyperRAB — A 20 IU/kg dose of Comparator HRIG will be given on Day 0 via IM injection.
  Other Names: HRIG
  Arms: Comparator HyperRab + RabAvert
Biological: RabAvert — A 1.0 ml dose of active vaccine (2.5 IU/ml) will be given IM on 5 occasions: on Days 0, 3, 7, 14, and 28.
  Other Names: active rabies vaccine

SUMMARY:
A prospective, randomized, blinded, parallel-group, non-inferiority, phase II/III study of the safety and effectiveness of simulated post-exposure prophylaxis with BPL HRIG with co-administration of active rabies vaccine in healthy subjects.

DETAILED DESCRIPTION:
Each subject will undergo a total of 9 visits. Subjects' eligibility will be assessed at Screening, which can occur up to 28 days prior to dosing. Following a repeat eligibility check at Day 0, eligible subjects will be randomized and dosed with the randomized treatment (BPL HRIG + vaccine or Comparator HRIG + vaccine) on Day 0. Further assessments will be conducted on Days 3, 5, 7, 14, 28, 49 and the end of study assessment on Day 140. Vaccine will be administered on Day 0, 3, 7, 14 and 28.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to sign an informed consent form.
2. Healthy male or female subjects aged 18 - 75 years inclusive.
3. No previous exposure to rabies virus, rabies vaccine and/or rabies immunoglobulin.
4. No significant abnormalities in hematology, biochemistry, or urinalysis according to the Principal Investigator's judgment.
5. No significant abnormalities in ECG according to the Investigator's judgment.
6. Females of child-bearing potential (defined from the onset of menstruation to one-year post- menopause and not surgically sterilized) who are (or become) sexually active must agree to practice contraception by using a highly effective (>98%) method for the duration of the study.
7. Females of child-bearing potential (defined from the onset of menstruation to one-year post- menopause and not surgically sterilized) must have a negative result on a serum at screening visit and a urine HCG-based pregnancy test at Day 0.

Exclusion Criteria

1. Female subjects who are pregnant and/or lactating.
2. History of live virus vaccination, e.g., measles, mumps, varicella or rubella vaccine, within the last 3 months.
3. Planned live virus vaccination, e.g., measles, mumps, varicella or rubella vaccine, within the 3 months after Day 0.
4. History of anaphylactic or anaphylactoid hypersensitivity reactions to chicken egg; history of mild allergic reactions to chicken egg, e.g., skin rash only, is not an exclusion criterion
5. History of hypersensitivity reaction to any of the following components of active rabies vaccine (US-FDA approved) e.g.: neomycin, bovine gelatin, trace amounts of chicken protein, chlortetracycline, and amphotericin B and in accordance with the product insert of the vaccine.
6. History of life-threatening allergy, anaphylactic reaction, or systemic response to human plasma derived products.
7. History of life-threatening allergy to blood or blood products.
8. Fever at the time of the start of the injection (oral temperature >38ºC.) or acute illness at the time of the start of the injection. Subjects with fever on Day 0 may have entry to the study re-scheduled.
9. History of or ongoing bleeding disorder.
10. Previous organ transplant recipient.
11. Ongoing immunosuppressive illness.
12. Clinically significant illnesses including: cardiac, hepatic, renal, endocrine, neurological, hematological, neoplastic, immunological, skeletal or other) that in the opinion of the investigator, could interfere with the safety, compliance or other aspects of this study.
13. All types of malignancies except for basal and squamous cell (scaly or plate-like) skin cancer, in- situ cervical carcinoma must be in remission for a minimum of 5 years prior to Day 0. For non-melanoma skin cancers and carcinoma in-situ of the cervix may be enrolled if treated and cured at the time of screening.
14. Evidence of active systemic infection that requires treatment with antibiotics within 2 weeks prior to Day 0.
15. Currently receiving or have received within the past 6 months (prior to Day 0):

    * immunosuppressive drugs
    * immunomodulatory drugs
16. Currently receiving or have received oral or IV steroids within 14 days (prior to DAY 0) or expected to require oral or IV steroids during the study.
17. Evidence of uncontrolled hypertension (systolic blood pressure of >150 mmHg, and/or diastolic blood pressure of >100 mmHg).
18. Heart rate >120/min.
19. Weight > 95.5 kg
20. History of IgA deficiency.
21. Is positive for any of the following at screening: serological test for HIV 1&2, HCV or HBsAg.
22. Presence of psychiatric disorder, other mental disorder or any other medical disorder which might impair the subject's ability to give informed consent or to comply with the requirements of the study protocol.
23. Previous enrollment in this study.
24. Participation in an interventional clinical trial within 30 days prior to baseline visit (Day 0).
25. Evidence of alcohol abuse or history of alcohol abuse or illegal and/or legally prescribed drugs in the past 2 years.
26. Any other factor that, in the opinion of the investigator, would prevent the subject from complying with the requirements of the protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2017-12-08 (Actual); Primary Completion 2018-03-02 (Actual); Study Completion 2018-07-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Holmes, MD, Study Director — Bio Products Laboratory
Locations (2):
- United States (2):
  - Prism Research, Saint Paul, Minnesota
  - Wake Research Associates, Raleigh, North Carolina

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BPL HRIG + RabAvert | Comparator HyperRab + RabAvert
Started | 81 | 81
Completed | 68 | 74
Not Completed | 13 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BPL HRIG + RabAvert | Comparator HyperRab + RabAvert | Total
Number analyzed (Participants) | 81 | 81 | 162
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.37 (15.0) | 44.56 (15.4) | 42.96 (15.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 54 | 110
  Male | 25 | 27 | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 79 | 78 | 157
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 16 | 15 | 31
  White | 62 | 59 | 121
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 81 | 81 | 162
Weight [Mean (Standard Deviation); unit: kg] | 74.61 (12.5) | 74.51 (13.2) | 74.56 (12.8)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects With Anti-rabies Antibody Titer of ≥0.5 IU/mL
Description: Non-inferiority in terms of the proportion of subjects with anti-rabies antibody titer of ≥0.5 IU/mL after study drug administration using a non-inferiority margin of 10%.
Time Frame: Day 14
Population: Primary PK population (all subjects who receive the full dose of BPL HRIG or comparator HRIG and the first 3 doses of active rabies vaccine on Days 0, 3, 7 and for whom the PK sample at Day 14 is taken).
Measure: Count of Participants; unit: Participants
Arm/Group | BPL HRIG + RabAvert | Comparator HyperRab + RabAvert
Number analyzed (Participants) | 73 | 74
Participants | 73 | 72
Statistical Analysis 1: Comparison: BPL HRIG + RabAvert vs Comparator HyperRab + RabAvert; Test type: Non-Inferiority — The null hypothesis is p-p0 ≤ -0.1. The alternative hypothesis is p-p0 > -0.1, where p is the proportion of subjects with anti-rabies titer of >0.5 IU/mL at Day 14 in subjects receiving BPL HRIG + vaccine and p0 is the proportion receiving comparator HRIG + vaccine. We reject the null hypothesis at the one-sided 0.025 significance level, and conclude that p-p0 > -0.1, if the lower bound of an exact 95% binomial confidence interval exceeds -0.1; p = 0.0006, Farrington and Manning test — The threshold for this test is <=0.025; lower 95% CI = -0.05, 95% CI 1-sided [lower limit -0.05]

2. Secondary Outcome: Analysis of AUC0-7d
Description: The AUC0-7d for BPL HRIG and vaccine versus comparator HRIG and vaccine using a non inferiority margin of 20%.
Time Frame: Day 0 to Day 7
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: day*IU/mL
Arm/Group | BPL HRIG + RabAvert | Comparator HyperRab + RabAvert
Number analyzed (Participants) | 73 | 74
day*IU/mL | 1.10 [1.02 to 1.20] | 1.32 [1.21 to 1.44]
Statistical Analysis 1: Comparison: BPL HRIG + RabAvert vs Comparator HyperRab + RabAvert; Test type: Non-Inferiority — The prespecified non inferiority margin was 20%. The lower bound of the 95% CI required should be greater than 0.8 to conclude non-inferiority; lower 95% CI = 0.74, 95% CI 2-sided [0.74 to 0.94]

3. Secondary Outcome: RVNA Geometric Mean Titers at Days 3, 5, 7 and 14
Description: Comparison of the geometric mean titers (GMTs) for antirabies antibody titer after administration of BPL HRIG and vaccine versus comparator HRIG and vaccine. The median peak RVNA titer occurred at Day 14, which is reflected in the analysis. The RVNA titer to peak geometric mean is analyzed using a repeated measures analysis. The inferential test compares RVNA values between BPL HRIG and HyperRab in a single analysis across all visits at or below the visit at which peak titer is observed. The geometric mean values presented represent a mean across all visits from baseline through and including Day 14.
Time Frame: Days 3, 5, 7 and 14
Population: Secondary PK population (subjects who receive the full dose of BPL HRIG or comparator HRIG and all 5 doses of active rabies vaccine and for whom all required PK samples are taken).
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | BPL HRIG + RabAvert | Comparator HyperRab + RabAvert
Number analyzed (Participants) | 61 | 69
IU/mL
  Through Day 14 | 0.37 [0.35 to 0.39] | 0.38 [0.36 to 0.40]
  Day 3 | 0.18 [0.16 to 0.20] | 0.21 [0.19 to 0.24]
  Day 5 | 0.19 [0.18 to 0.21] | 0.24 [0.21 to 0.26]
  Day 7 | 0.23 [0.21 to 0.26] | 0.26 [0.23 to 0.29]
  Day 14 | 12.30 [10.15 to 14.90] | 8.38 [6.54 to 10.74]
Statistical Analysis 1: Comparison: BPL HRIG + RabAvert vs Comparator HyperRab + RabAvert; Test type: Superiority; 95% CI = 0.97 — Data analyzed as log normal. The value presented is the untransformed value of the difference between means

4. Secondary Outcome: Proportion of Subjects Reaching Antirabies Antibody Titer of ≥ 0.5 IU/mL by Visit
Description: The proportion of subjects reaching antirabies antibody titer of ≥ 0.5 IU/mL after administration of BPL HRIG and vaccine versus comparator HRIG and vaccine.
Time Frame: Days 3, 5, 7, 14, 28, 49, and 140
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BPL HRIG + RabAvert | Comparator HyperRab + RabAvert
Number analyzed (Participants) | 73 | 74
Participants
  Day 0 | 0 | 0
  Day 3 | 0 | 1
  Day 5: number analyzed (Participants) | 71 | 74
  Day 5 | 0 | 1
  Day 7 | 3 | 2
  Day 14 | 73 | 72
  Day 28 | 73 | 73
  Day 49: number analyzed (Participants) | 73 | 72
  Day 49 | 73 | 72
  Day 140: number analyzed (Participants) | 62 | 71
  Day 140 | 60 | 65
Statistical Analysis 1: Comparison: BPL HRIG + RabAvert vs Comparator HyperRab + RabAvert; Test type: Non-Inferiority — The same methodology was used as the primary endpoint for each visit. The statistical analysis is presenting the Day 14 data; p = 0.0006, Farrington and Manning test; lower 95% CI = -0.05, 95% CI 2-sided [-0.05 to 0.10]

5. Secondary Outcome: Proportion of Subjects Reaching Antirabies Antibody Titer of ≥ LLOQ of the Assay by Visit
Description: The proportion of subjects reaching antirabies antibody titer of ≥ LLOQ of the assay at each visit after administration of BPL HRIG and vaccine versus comparator HRIG and vaccine.
Time Frame: Days 3, 5, 7, 14, 28, 49, and 140
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BPL HRIG + RabAvert | Comparator HyperRab + RabAvert
Number analyzed (Participants) | 73 | 74
Participants
  Day 0 | 0 | 0
  Day 3 | 70 | 73
  Day 5: number analyzed (Participants) | 71 | 74
  Day 5 | 71 | 74
  Day 7 | 73 | 74
  Day 14 | 73 | 74
  Day 28 | 73 | 74
  Day 49: number analyzed (Participants) | 73 | 72
  Day 49 | 73 | 72
  Day 140: number analyzed (Participants) | 62 | 71
  Day 140 | 62 | 71
Statistical Analysis 1: Comparison: BPL HRIG + RabAvert vs Comparator HyperRab + RabAvert; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p = 0, Farrington and Manning test; lower 95% CI = 0, 95% CI 2-sided [0 to 0] — For Day 14, all subjects achieved the endpoint (RVNA titer > LLOQ). Since the statistic to measure the performance is a proportion, the proportion is 1 and no variance is calculable

6. Secondary Outcome: RVNA Geometric Mean Titers at Days 14, 28, 49 and 140
Description: Comparison of the GMTs for antirabies antibody titer after administration of BPL HRIG and vaccine versus comparator HRIG and vaccine to assess the inhibitory effects of BPL HRIG on active immunization relative to that of the comparator HRIG.
Time Frame: Days 14, 28, 49 and 140
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | BPL HRIG + RabAvert | Comparator HyperRab + RabAvert
Number analyzed (Participants) | 61 | 69
IU/mL
  Day 14 | 12.30 [10.15 to 14.90] | 8.38 [6.54 to 10.74]
  Day 28 | 10.18 [8.39 to 12.34] | 7.78 [6.26 to 9.66]
  Day 49 | 10.91 [8.94 to 13.32] | 7.78 [6.34 to 9.56]
  Day 140 | 2.72 [2.21 to 3.34] | 2.02 [1.62 to 2.53]

ADVERSE EVENTS:
Time Frame: 20 weeks treatment
Description: Includes treatment emergent adverse events
Arm/Group | BPL HRIG + RabAvert | Comparator HyperRab + RabAvert
All-Cause Mortality (participants affected / at risk) | 0/81 | 0/81
Serious Adverse Events (participants affected / at risk) | 0/81 | 0/81
Other Adverse Events (participants affected / at risk) | 19/81 | 19/81
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BPL HRIG + RabAvert (N=81) | Comparator HyperRab + RabAvert (N=81)
Vaccination site pain (General disorders) | 9 (10) | 2 (3) — Vaccination site pain AEs were related to the vaccine dose administration.
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 7 (7)
Headache (Nervous system disorders) | 5 (5) | 10 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2017-10-26): https://cdn.clinicaltrials.gov/large-docs/57/NCT03264157/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-31): https://cdn.clinicaltrials.gov/large-docs/57/NCT03264157/SAP_001.pdf